CLINICAL TRIAL: NCT01659593
Title: Evaluation of the Efficiency of a Cognitive Remedial Program (PROCOG-SEP) Designed for Multiple Sclerosis Patients. A Double Blind Randomized Multicenter Trial.
Brief Title: Evaluation of the Efficiency of a Cognitive Remedial Program (PROCOG-SEP) Designed for Multiple Sclerosis Patients
Acronym: PROCOG-SEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: University Hospital, Strasbourg, France (Other); Centre Hospitalier Universitaire Dijon (Other); Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROCOG-SEP
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Cognitive Disorders; Multiple Sclerosis
Keywords: cognitive disorders; multiple sclerosis; neuropsychology
MeSH Terms: conditions — Cognitive Dysfunction; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- procog (Experimental): cognitive remedial program 13 sessions over a 6-month period
  Interventions: Other: procog
- DISINT (Placebo Comparator): Interactive discussion program of 13 group sessions in a 6-month period
  Interventions: Other: Placebo

INTERVENTIONS:
Other: procog — 3 to 5 people group program
  Arms: procog
Other: Placebo
  Arms: DISINT

SUMMARY:
Cognitive disorders are well-known in multiple sclerosis (MS), even in earlier stages of the disease. They effect personal life. Their management may be overlooked. The evidence-based program proposes exercises to both stimulate preserved functions and develop new abilities compensating for cognitive disabilities.

Aim of the study is to evaluate the efficiency of the remedial program (PROCOG-SEP) designed for MS patients, compared to an interactive discussion program(DISINT) 140 multiple sclerosis patients will be randomly assigned in one the program for 13 sessions over a 6-month period.

Main outcome criteria is evolution of SRT-LIST before and after program.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤Aged ≤ 60 at baseline
* Must be able to understand and read french language
* Must sign the informed consent form
* Must be affiliate to French social security
* multiple sclerosis confirmed by Mac Donald criteria
* EDSS ≤ 6.0 at baseline
* Duration of multiple sclerosis ≤ 30 years at baseline
* mild cognitive disorder ( at least 2 cognitive tasks, at most 5 )

Exclusion Criteria:

* under legal protection
* treatment by corticosteroids in the past 4 weeks
* cognitive remedial program already done
* neuropsychologic assessment in the past 2 months
* having an other chronic disease
* having an other neurologic disease
* alcohol or drug addiction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-09 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
cognitive function measured by SRT-List score | 0-9 months

SECONDARY OUTCOMES:
quality of life measured by MusiQol | 0 -9 months

OTHER OUTCOMES:
cognitive function: verbal memory (SRT), visuospatial memory (10/36), verbal fluency (animal categories),empans, code ,DO80, cognitive complaint | 0-9 months

CONTACTS AND LOCATIONS:
Overall Officials: Marc DEBOUVERIE, Professor, Principal Investigator — CHU NANCY; Eric BERGER, MD, Principal Investigator — CHU DE BESANCON; Thibaut MOREAU, Professor, Principal Investigator — Centre Hospitalier Universitaire Dijon; Jérôme de Sèze, Professor, Principal Investigator — CHU de STRASBOURG
Locations (1):
- University hospital Nancy, Nancy, France